CLINICAL TRIAL: NCT03576066
Title: A Phase 2a, Multi-center, Double-blind, Placebo-controlled Study Evaluating ABI-H0731 as Adjunctive Therapy in Virally-suppressed Patients With Chronic Hepatitis B
Brief Title: A Study Evaluating ABI-H0731 as Adjunctive Therapy in Participants With Chronic Hepatitis B Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assembly Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ABI-H0731-201
Record Dates: First submitted 2018-06-06; First posted 2018-07-03 (Actual); Results first posted 2021-01-28 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-01

CONDITIONS: Chronic Hepatitis B
Keywords: Chronic hepatitis B; HBV; HBeAg-positive; hepatitis B; HBeAg-negative; vebicorvir; VBR
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B | interventions — entecavir; Tenofovir; tenofovir alafenamide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ABI-H0731 + SOC NUC (Experimental): Virologically suppressed participants will receive ABI-H0731 along with SOC NUC (ETV, TDF or TAF) tablets orally for 24 weeks. Eligible participants may enter a separate extension study after Week 24 to continue open-label ABI-H0731 for up to an additional year if necessary.
  Interventions: Drug: ABI-H0731; Drug: SOC NUC
- Placebo + SOC NUC (Active Comparator): Virologically suppressed participants will receive matching placebo tablets and continue their SOC NUC (ETV, TDF or TAF) for 24 weeks. Eligible participants may enter a separate extension study after Week 24 to start treatment on open-label ABI-H0731 for up to a year if necessary.
  Interventions: Drug: SOC NUC; Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: ABI-H0731 — Participants will receive ABI-H0731 300 mg tablets orally once daily (QD).
  Arms: ABI-H0731 + SOC NUC
Drug: SOC NUC — Participants will continue on their SOC NUC (ETV, TDF or TAF) tablet orally as per approved package insert.
  Other Names: Entecavir (ETV); Tenofovir disoproxil fumarate (TDF); Tenofovir alafenamide (TAF)
Drug: Placebo Oral Tablet — Participants will receive placebo matching ABI-0731 tablets orally QD.
  Arms: Placebo + SOC NUC

SUMMARY:
The purpose of this study is to determine if ABI-H0731 given in combination with a standard of care (SOC) hepatitis B virus (HBV) nucleos(t)ide reverse transcriptase inhibitor (NUC) medication is safe and effective in participants with chronic hepatitis B virus infection (cHBV).

DETAILED DESCRIPTION:
This is a Phase 2a, Multi-center, Double-blind, Placebo-controlled Study Evaluating ABI-H0731 as Adjunctive Therapy in Virally-suppressed Participants with cHBV.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female between ages 18 and 70 years
* Virologically-suppressed (defined as HBV DNA ≤limit of quantitation (LOQ) for at least 6 months before screening on SOC NUC therapy
* HBeAg-positive or HBeAg-negative at screening
* In good general health except for cHBV

Key Exclusion Criteria:

* Co-infection with HIV, hepatitis C virus (HCV), hepatitis E virus (HEV) or hepatitis D virus (HDV)
* History or evidence of hepatic decompensation (including gastrointestinal bleeding or esophageal varices) at any time prior to or at time of screening
* Clinically significant cardiac or pulmonary disease, chronic or recurrent renal or urinary tract disease, liver disease other than HBV, endocrine disorder, autoimmune disorder, diabetes mellitus requiring treatment with insulin or hypoglycemic agents, neuromuscular, musculoskeletal, or mucocutaneous conditions requiring frequent treatment, seizure disorders requiring treatment, or other medical conditions requiring frequent medical management or pharmacologic or surgical treatment that in the opinion of the Investigator or the Sponsor makes the participant unsuitable for the study
* Previous treatment with an investigational agent for HBV other than ABI-H0731 in the last 6 months before screening
* History of hepatocellular carcinoma (HCC)
* Females who are lactating or pregnant or wish to become pregnant are excluded from the study
* Exclusionary laboratory parameters at screening include:

  * Platelet count <100,000/mm3
  * Albumin <lower limit of normal (LLN)
  * Direct bilirubin >1.2×upper limit of normal (ULN)
  * Alanine aminotransferase (ALT) >5×ULN at screening
  * International Normalized Ratio (INR) >1.5×ULN
  * Glomerular filtration rate (GFR) <60 mL/min/1.73 m2 by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2019-07-05 (Actual); Study Completion 2019-07-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (21):
- United States (17):
  - Cedars-Sinai Medical Center, Beverly Hills, California
  - Southern California Research Center, Coronado, California
  - Asia Pacific Liver Center, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - Research and Education, San Diego, California
  - Medical Associates Research Group, San Diego, California
  - Quest Clinical Research, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - University of Miami Hospital and Clinics, Miami, Florida
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Digestive Disease Associates, Catonsville, Maryland
  - Infectious Disease Care, Hillsborough, New Jersey
  - Sing Chan, MD, Flushing, New York
  - NYU Langone Health, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Xiaoli Ma, MD, Philadelphia, Pennsylvania
- Canada (3):
  - Toronto General Hospital, Toronto
  - Toronto Liver Center, Toronto
  - GI Research Institute, Vancouver
- Auckland City Hospital, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yuen MF, Agarwal K, Ma X, Nguyen TT, Schiff ER, Hann HL, Dieterich DT, Nahass RG, Park JS, Chan S, Han SB, Gane EJ, Bennett M, Alves K, Evanchik M, Yan R, Huang Q, Lopatin U, Colonno R, Ma J, Knox SJ, Stamm LM, Bonacini M, Jacobson IM, Ayoub WS, Weilert F, Ravendhran N, Ramji A, Kwo PY, Elkhashab M, Hassanein T, Bae HS, Lalezari JP, Fung SK, Sulkowski MS. Safety and efficacy of vebicorvir in virologically suppressed patients with chronic hepatitis B virus infection. J Hepatol. 2022 Sep;77(3):642-652. doi: 10.1016/j.jhep.2022.04.005. Epub 2022 Apr 20. PMID 35460726

RESULTS

PARTICIPANT FLOW:
Groups:
- ABI-H0731 + SOC NUC: Virologically suppressed participants will receive ABI-H0731 along with standard of care (SOC) nucleos(t)ide reverse transcriptase inhibitor (NUC) tablets orally for 24 weeks. Eligible participants may enter a separate extension study after Week 24 to continue open-label ABI-H0731 for up to an additional year if necessary.
  ABI-H0731: Participants will receive 300 mg QD ABI-H0731 tablets orally.
  SOC NUC: Participants will continue on their SOC NUC (ETV, TDF or TAF) tablet orally (QD frequency) as per approved package insert.
- Placebo + SOC NUC: Virologically suppressed participants will receive matching placebo tablets and continue their SOC NUC (ETV, TDF or TAF) for 24 weeks. Eligible participants may enter a separate extension study after Week 24 to start treatment on open-label ABI-H0731 for up to a year if necessary.
  Placebo Oral Tablet: Participants will receive matching QD placebo tablets orally.
  SOC NUC: Participants will receive SOC NUC (ETV, TDF or TAF) tablet orally as per approved package insert.
Period: Overall Study
Arm/Group | ABI-H0731 + SOC NUC | Placebo + SOC NUC
Started | 45 | 28
Completed | 45 | 27
Not Completed | 0 | 1
Not completed — Noncompliance with study drug | 0 | 1

BASELINE CHARACTERISTICS:
Population: Randomized participants
Groups:
- ABI-H0731 + SOC NUC: Virologically suppressed participants will receive ABI-H0731 along with SOC NUC (ETV, TDF or TAF) tablets orally for 24 weeks. Eligible participants may enter a separate extension study after Week 24 to continue open-label ABI-H0731 for up to an additional year if necessary.
  ABI-H0731: Participants will receive 300 mg QD ABI-H0731 tablets orally.
  SOC NUC: Participants will continue on their SOC NUC (ETV, TDF or TAF) tablet orally (QD frequency) as per approved package insert.
- Total: Total of all reporting groups
Arm/Group | ABI-H0731 + SOC NUC | Placebo + SOC NUC | Total
Number analyzed (Participants) | 45 | 28 | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.6 (10.26) | 46.4 (11.32) | 45.3 (10.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 32 | 15 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 44 | 27 | 71
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 37 | 24 | 61
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 2 | 3 | 5
  White | 4 | 0 | 4
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  New Zealand | 1 | 0 | 1
  Canada | 6 | 4 | 10
  United States | 37 | 24 | 61
  Hong Kong | 1 | 0 | 1
Hepatitis B "e" Antigen (HBeAg) status [Count of Participants; unit: Participants]
  HBeAg Positive | 29 | 18 | 47
  HBeAg Negative | 16 | 10 | 26

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean log10 Serum HBsAg From Baseline (Day 1) to Week 24 on ABI-H0731 + SOC NUC as Compared to Placebo + SOC NUC
Time Frame: Baseline to Week 24
Population: Intention-to-treat (ITT) population: all randomized participants. Results were analyzed and reported based on Baseline HBeAg status: positive or negative, for available data at Baseline, Week 24, or both.
Measure: Mean (Standard Deviation); unit: Log10 International Units (IU)/mL
Groups:
- HBeAg-positive Participants: ABI-H0731 + SOC NUC: Virologically suppressed participants who are HBeAg positive at Baseline will receive ABI-H0731 along with SOC NUC (ETV, TDF or TAF) tablets orally for 24 weeks. Eligible participants may enter a separate extension study after Week 24 to continue open-label ABI-H0731 for up to an additional year if necessary.
  ABI-H0731: Participants will receive 300 mg QD ABI-H0731 tablets orally.
  SOC NUC: Participants will continue on their SOC NUC (ETV, TDF or TAF) tablet orally (QD frequency) as per approved package insert.
- HBeAg-positive Participants: Placebo + SOC NUC: Virologically suppressed participants who are HBeAg positive at Baseline will receive matching placebo tablets and continue their SOC NUC (ETV, TDF or TAF) for 24 weeks. Eligible participants may enter a separate extension study after Week 24 to start treatment on open-label ABI-H0731 for up to a year if necessary.
  Placebo Oral Tablet: Participants will receive matching QD placebo tablets orally.
  SOC NUC: Participants will receive SOC NUC (ETV, TDF or TAF) tablet orally as per approved package insert.
- HBeAg-negative Participants: ABI-H0731 + SOC NUC: Virologically suppressed participants who are HBeAg negative at Baseline will receive ABI-H0731 along with SOC NUC (ETV, TDF or TAF) tablets orally for 24 weeks. Eligible participants may enter a separate extension study after Week 24 to continue open-label ABI-H0731 for up to an additional year if necessary.
  ABI-H0731: Participants will receive 300 mg QD ABI-H0731 tablets orally.
  SOC NUC: Participants will continue on their SOC NUC (ETV, TDF or TAF) tablet orally (QD frequency) as per approved package insert.
- HBeAg-negative Participants: Placebo + SOC NUC: Virologically suppressed participants who are HBeAg negative at Baseline will receive matching placebo tablets and continue their SOC NUC (ETV, TDF or TAF) for 24 weeks. Eligible participants may enter a separate extension study after Week 24 to start treatment on open-label ABI-H0731 for up to a year if necessary.
  Placebo Oral Tablet: Participants will receive matching QD placebo tablets orally.
  SOC NUC: Participants will receive SOC NUC (ETV, TDF or TAF) tablet orally as per approved package insert.
Arm/Group | HBeAg-positive Participants: ABI-H0731 + SOC NUC | HBeAg-positive Participants: Placebo + SOC NUC | HBeAg-negative Participants: ABI-H0731 + SOC NUC | HBeAg-negative Participants: Placebo + SOC NUC
Number analyzed (Participants) | 29 | 18 | 16 | 10
Log10 International Units (IU)/mL
  Baseline | 3.48 (0.401) | 3.57 (0.516) | 2.99 (0.555) | 3.35 (0.648)
  Change from baseline: number analyzed (Participants) | 29 | 17 | 16 | 10
  Change from baseline | 0.03 (0.138) | 0.03 (0.054) | 0.09 (0.133) | -0.00 (0.021)
Statistical Analysis 1: Comparison: HBeAg-positive Participants: ABI-H0731 + SOC NUC vs HBeAg-positive Participants: Placebo + SOC NUC; Least squares (LS) mean difference in HBeAg-positive participants: ABI-H0731 + SOC NUC minus placebo + SOC NUC at Week 24; Test type: Other; p = 0.6855, Repeated measures analysis
Statistical Analysis 2: Comparison: HBeAg-negative Participants: ABI-H0731 + SOC NUC vs HBeAg-negative Participants: Placebo + SOC NUC; LS mean difference in HBeAg-negative participants: ABI-H0731 + SOC NUC minus placebo + SOC NUC at Week 24; Test type: Other; p = 0.1750, Repeated measures analysis

2. Primary Outcome: Change in Mean log10 Serum HBeAg From Baseline (Day 1) to Week 24 on ABI-H0731 + SOC NUC as Compared to Placebo + SOC NUC
Time Frame: Baseline to Week 24
Population: ITT population. Results were analyzed and reported only for participants who were HBeAg positive at Baseline and had available data at Baseline, Week 24, or both.
Measure: Mean (Standard Deviation); unit: Log10 International Units (IU)/mL
Arm/Group | HBeAg-positive Participants: ABI-H0731 + SOC NUC | HBeAg-positive Participants: Placebo + SOC NUC
Number analyzed (Participants) | 29 | 18
Log10 International Units (IU)/mL
  Baseline | 0.55 (0.980) | 0.43 (0.964)
  Change from baseline: number analyzed (Participants) | 29 | 16
  Change from baseline | -0.05 (0.191) | -0.10 (0.193)
Statistical Analysis 1: Comparison: HBeAg-positive Participants: ABI-H0731 + SOC NUC vs HBeAg-positive Participants: Placebo + SOC NUC; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.2916, Repeated measures analysis

3. Secondary Outcome: Number of Participants With One or More Adverse Events
Time Frame: Up to Follow-up (maximum up to Week 36)
Population: Safety population: all randomized participants who received any amount of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | ABI-H0731 + SOC NUC | Placebo + SOC NUC
Number analyzed (Participants) | 45 | 28
Participants | 24 | 8

4. Secondary Outcome: Number of Participants With Premature Study Discontinuation
Time Frame: Up to Follow-up (maximum up to Week 36)
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | ABI-H0731 + SOC NUC | Placebo + SOC NUC
Number analyzed (Participants) | 45 | 28
Participants | 0 | 1

5. Secondary Outcome: Number of Participants With One or More Abnormal Safety Laboratory Result
Time Frame: Up to Week 36
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | ABI-H0731 + SOC NUC | Placebo + SOC NUC
Number analyzed (Participants) | 45 | 28
Participants | 27 | 20

6. Secondary Outcome: Number of Participants With a Clinically-significant Electrocardiogram Abnormality
Time Frame: Up to Week 24
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | ABI-H0731 + SOC NUC | Placebo + SOC NUC
Number analyzed (Participants) | 45 | 28
Participants | 0 | 0

7. Secondary Outcome: Number of Participants With a Clinically-significant Change in Vital Signs
Description: Vital signs assessed were body temperature, respiratory rate, and pulse rate
Time Frame: Baseline and up to Week 24
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | ABI-H0731 + SOC NUC | Placebo + SOC NUC
Number analyzed (Participants) | 45 | 28
Participants | 0 | 0

8. Secondary Outcome: Number of Participants With Abnormal Alanine Aminotransferase (ALT) at Baseline Who Have Normal ALT at Week 24 on ABI-H0731 + NUC Therapy as Compared With Placebo + NUC Therapy
Description: Abnormal ALT was defined as ≥1.25 x upper limit of normal (34 Units/L for female and 43 Units/L for male participants).
Time Frame: Baseline to Week 24
Population: Participants in the ITT population with abnormal ALT at Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | ABI-H0731 + SOC NUC | Placebo + SOC NUC
Number analyzed (Participants) | 2 | 1
Participants | 1 | 0

9. Secondary Outcome: Trough Levels of ABI-H0731 on ABI-H0731 + SOC NUC Therapy
Time Frame: Before dosing at Baseline (Day 1), Weeks 2, 4, 12, and 24
Population: Safety population. Results were analyzed and reported only for participants who received ABI-H0731 + SOC NUC and had ABI-H0731 pharmacokinetic data assessments available.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ABI-H0731 + SOC NUC
Number analyzed (Participants) | 45
ng/mL
  Baseline (Day 1) | 0.436 (2.92)
  Week 2 | 1390 (647)
  Week 4: number analyzed (Participants) | 44
  Week 4 | 1390 (632)
  Week 12 | 1330 (560)
  Week 24 | 1330 (526)

10. Secondary Outcome: Trough Levels of Entecavir (ETV) on ABI-H0731 + SOC NUC Therapy as Compared With Placebo + SOC NUC Therapy
Time Frame: Before dosing at Baseline (Day 1), Weeks 2, 4, 12, and 24
Population: Safety population. Results were analyzed and reported only for participants who received ETV as their SOC NUC and had ETV pharmacokinetic data assessments available.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ABI-H0731 + SOC NUC | Placebo + SOC NUC
Number analyzed (Participants) | 7 | 3
ng/mL
  Baseline (Day 1) | 1.10 (1.88) | 1.78 (1.77)
  Week 2 | 0.554 (0.261) | 0.346 (0.124)
  Week 4 | 0.872 (1.04) | 0.621 (0.460)
  Week 12: number analyzed (Participants) | 7 | 2
  Week 12 | 0.583 (0.363) | 0.704 (0.403)
  Week 24 | 1.04 (1.57) | 0.739 (0.0902)

11. Secondary Outcome: Trough Levels of Tenofovir Alafenamide (TAF) on ABI-H0731 + SOC NUC Therapy as Compared With Placebo + SOC NUC Therapy
Time Frame: Before dosing at Baseline (Day 1), Weeks 2, 4, 12, and 24
Population: Safety population. Results were analyzed and reported only for participants who received TAF as their SOC NUC and had TAF pharmacokinetic data assessments available.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ABI-H0731 + SOC NUC | Placebo + SOC NUC
Number analyzed (Participants) | 14 | 8
ng/mL
  Baseline (Day 1) | 9.67 (3.43) | 12.2 (6.52)
  Week 2 | 13.1 (4.73) | 14.1 (6.95)
  Week 4: number analyzed (Participants) | 13 | 8
  Week 4 | 21.3 (25.3) | 11.8 (4.52)
  Week 12 | 18.4 (14.3) | 11.7 (3.66)
  Week 24 | 18.9 (18.2) | 13.3 (3.26)

12. Secondary Outcome: Trough Levels of Tenofovir Disoproxil Fumarate (TDF) on ABI-H0731 + SOC NUC Therapy as Compared With Placebo + SOC NUC Therapy
Time Frame: Before dosing at Baseline (Day 1), Weeks 2, 4, 12, and 24
Population: Safety population. Results were analyzed and reported only for participants who received TDF as their SOC NUC and had TDF pharmacokinetic data assessments available.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ABI-H0731 + SOC NUC | Placebo + SOC NUC
Number analyzed (Participants) | 23 | 15
ng/mL
  Baseline (Day 1) | 77.5 (52.1) | 89.1 (71.4)
  Week 2 | 85.5 (49.3) | 76.2 (21.5)
  Week 4: number analyzed (Participants) | 23 | 14
  Week 4 | 86.8 (58.2) | 84.1 (60.3)
  Week 12: number analyzed (Participants) | 20 | 15
  Week 12 | 79.3 (68.1) | 86.7 (47.4)
  Week 24 | 79.3 (45.3) | 78.3 (44.4)

13. Secondary Outcome: Trough to Peak Ratios of ABI-H0731 on ABI-H0731 + SOC NUC Therapy
Time Frame: Baseline, Weeks 2, 4, 12, and 24
Population: Trough to peak ratios were not calculated due to an insufficient number of optional peak exposure samples.
Arm/Group | ABI-H0731 + SOC NUC
Number analyzed (Participants) | 0

14. Secondary Outcome: Trough to Peak Ratios of SOC NUC on ABI-H0731 + SOC NUC Therapy as Compared With Placebo + SOC NUC Therapy
Time Frame: Baseline, Weeks 2, 4, 12, and 24
Population: Trough to peak ratios were not calculated due to an insufficient number of optional peak exposure samples.
Arm/Group | ABI-H0731 + SOC NUC | Placebo + SOC NUC
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to Week 36
Description: Safety population
Arm/Group | ABI-H0731 + SOC NUC | Placebo + SOC NUC
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/28
Other Adverse Events (participants affected / at risk) | 24/45 | 8/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABI-H0731 + SOC NUC (N=45) | Placebo + SOC NUC (N=28)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Influenza (Infections and infestations) | 2 (2) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Bacterial vaginosis (Infections and infestations) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Onychomycosis (Infections and infestations) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tongue ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (2)
Fatigue (General disorders) | 1 (1) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Inflammation (General disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hepatic pain (Hepatobiliary disorders) | 1 (1) | 0 (0)
Liver tenderness (Hepatobiliary disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0)
Libido decreased (Psychiatric disorders) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Assembly Biosciences agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Assembly Biosciences supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-11-09): https://cdn.clinicaltrials.gov/large-docs/66/NCT03576066/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-06): https://cdn.clinicaltrials.gov/large-docs/66/NCT03576066/SAP_001.pdf